CLINICAL TRIAL: NCT04136665
Title: Physical Activity Adapted at Home Supervised by Videoconferencing in Post-cancer for Children / AYA Treated for Leukemia: Reduction of Territorial and Social Inequalities Due to E-health - Feasibility Study (ONCOPED SAPATIC)
Brief Title: Physical Activity Adapted at Home Supervised by Videoconferencing in Post-cancer for Children / AYA Treated for Leukemia (ONCOPED SAPATIC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patient
Sponsor: University Hospital, Montpellier (Other)
Collaborators: mooven society (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL19_0181
Record Dates: First submitted 2019-10-18; First posted 2019-10-23 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-01

CONDITIONS: Leukemia
Keywords: children; leukemia; physical activity adapted
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity Adapted program (Experimental)
  Interventions: Other: Physical Activity Adapted program

INTERVENTIONS:
Other: Physical Activity Adapted program — 6-month APA home program, supervised by videoconferencing in post-cancer for children / AYA treated for leukemia

SUMMARY:
Leukemia is the most common form of cancer (29%) in children, adolescents, and young adults (AYA) (CNIB Report, 2017). Current treatments for leukemia (conventional chemotherapy or hematopoietic stem cell transplantation) can lead to significant side effects, acute or chronic, which can lead to impaired physical abilities and reduced quality of life for patients in short, medium or long term. For children and AYA with cancer, adapted physical activity (APA) is now recommended even if the scientific evidence of its benefit is still insufficient.

DETAILED DESCRIPTION:
Leukemia is the most common form of cancer (29%) in children, adolescents, and young adults (AYA). Current treatments for leukemia (conventional chemotherapy or hematopoietic stem cell transplantation) can lead to significant side effects, acute or chronic, which can lead to impaired physical abilities and reduced quality of life for patients in short, medium or long term. For children and AYA with cancer, adapted physical activity (APA) is now recommended even if the scientific evidence of its benefit is still insufficient. However, some publications show clearly the benefits of an APA program for this population. It is important to note that these studies (and therefore the evaluated APA programs) were carried out during hospitalization, where a significant sedentary situation was reported in children/AYA with cancer, especially on their return home. The main barriers to the practice of APA, recently described in the literature, are: 1 / Patient's distance from the health center (geographical and social inequality); 2 / Insufficient involvement of the family environment (social inequality); 3 / Social rupture of the child / AYA. To neutralize these particularly marked inequalities in post-cancer period, the introduction of a home-based APA program represents an innovative and relevant solution. Thus, it was reported that 91% (out of 1500 participants) of children / AYAs with cancer wish to engage in physical activity at home regardless the time of the care course. In addition, the use of new information and communication technologies (ICT) such as videoconferencing does not constitute a barrier to the practice of APA for this young population familiar with connected tools. The practice of APA could even be an important lever in the fight against sedentary lifestyle by inducing a long-term change in behavior. In order to achieve these objectives, the APA programs in children/AYA with cancer should meet 3 major criteria: 1 / Professionally supervised sessions; 2 / Progressive increase in number and intensity of sessions; 3 / Accompanying the patient to an independent practice of regular physical activity. To date, the studies reported in literature have proposed "APA follow-ups" at home only by mail, telephone or via internet applications. Their effects appear limited on physical capacities for children/AYAs with cancer. However, according to these authors, setting up a home-based APA program through the use of ICTs would maximize the benefits on the physical capabilities and quality of life of all these patients. To the investigator's knowledge, no study has yet been conducted to evaluate the feasibility of such a program, and its consequences on patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Leukemia and followed in intensive post-treatment or with lymphoma and followed in post autologous graft, patient aged 12 to 25 years old (child/AYA), included in the CHU Montpellier and identified by the mobile support team AYA Occitanie-Est, and or the Occitanie-Est Pediatric Division of the Oncology Network of the Occitanie Region,
* Having completed and signed a consent form for the study (Signature of consent by the parents if the patient is a minor)
* affiliated to a safety social regime

Exclusion Criteria:

* Contraindication to the practice of an APA program.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
evaluate the feasibility of a 6-month APA home program, supervised by videoconferencing in post-cancer for children / AYA treated for leukemia: number of completed session / number of theorical session | 6 months
  Assessment of the feasibility of a 6-month APA home program, supervised by videoconferencing in post-cancer for children / AYA treated for leukemia : number of completed session / number of theorical session

SECONDARY OUTCOMES:
evaluate the impact of a 6-month APA home program on the muscle strength of lower limbs | 6 months
  Assessment of the muscle strength of lower limbs by the 30s chair test at the beginning and at the end of the APA home program
evaluate the impact of a 6-month APA home program on the exercise capacity | 6 months
  Assessment of the exercise capacity by the six minutes walk test at the beginning and the end of the study
evaluate the impact of a 6-month APA home program on the muscle flexibility | 6 months
  Assessment of the muscle flexibility by the sit and reach test at the beginning and the end of the study
evaluate the impact of a 6-month APA home program on the quality of life: PedsQL | 6 months
  Assessment of the quality of life by the PedsQL at the beginning and the end of study

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Montpellier, Montpellier, France